CLINICAL TRIAL: NCT03980678
Title: Effect of Red Algae Lithothamnion on Blood Lactate Response During Exhaustive Exercise in Trained Cyclists: A Randomized Control Trial
Brief Title: Lithothamnion Species on Blood Lactate During Exhaustive Exercise in Trained Cyclists
Acronym: AAPt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAPtrial
Record Dates: First submitted 2019-05-28; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Exercise-Induced Lactic Acidemia; Lactate Blood Increase
Keywords: Mineral Rich Algae; Mineral Nutrition
MeSH Terms: conditions — Hyperlactatemia | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: One week (7 day) supplementation, followed by a 4 week washout, then crossover (another 7 day supplementation period).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties directly involved in recruitment, data collection and analysis will be blinded to the supplement identities until after the data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mineral Rich Algae with orange flavoring (Active Comparator): Participants will consume the Aquamin Soluble (Mineral Rich Algae) equivalent of 1000mg Calcium in 250 ml of orange flavoured water.
  Interventions: Dietary Supplement: Mineral Rich Algae
- Water with orange flavoring (Placebo Comparator): Participants will consume a placebo of maltodextrin in 250 ml of orange flavoured water (40mg Calcium).
  Interventions: Dietary Supplement: Orange flavoured water with maltodextrin as the placebo

INTERVENTIONS:
Dietary Supplement: Mineral Rich Algae — Lithothamnion species is rich in calcium, magnesium (Mg) and 72 other trace elements absorbed from sea-water during the organisms life. Mineral-rich 'fronds' break off from the living organism, fall to the ocean floor and are harvested (AquaminF). The mineral extract in soluble form contains ~13.1% Calcium, ~1.04% Magnesium and measurable levels of 72 other trace minerals. Following or prior to a washout period (crossover intervention), participants will consume the Aquamin Soluble equivalent of 1000mg Calcium in 250 ml of orange flavored water for a 7 day loading period.
  Other Names: Aquamin soluble
  Arms: Mineral Rich Algae with orange flavoring
Dietary Supplement: Orange flavoured water with maltodextrin as the placebo — Following or prior to a washout period (crossover intervention), participants will consume 250 ml of orange flavoured water (containing 20mg of Calcium with maltodextrin) for a 7 day period.
  Other Names: Placebo
  Arms: Water with orange flavoring

SUMMARY:
Deep ocean mineral water has been shown to improve exercise phenotypes in human and animal models. However, there is yet to be an investigation of Algae species such as Lithothamnion that absorb and concentrate these minerals. Therefore, the AAP trial will investigate the effect of water soluble Lithothamnion species on exhaustive exercise-induced blood lactate accumulation, recovery and power output in trained cyclists.

DETAILED DESCRIPTION:
The potential for naturally derived combinations of marine minerals to improve exercise performance is growing throughout the scientific literature and has physiologically plausible mechanisms, likely through the diverse molecular and enzymatic actions of individual (or combinations of) minerals (such as Calcium and Magnesium).

Despite the biological potential, there is little consciences whether mineral supplementation can improving markers of, and exercise performance. One recent investigation of deep ocean mineral water (high in marine minerals) showed that when consumed prior to exercise, blood lactate response improved with hyperthermal running and is supported in animal models - however, this is not supported elsewhere in humans. Nonetheless, others have shown, in human models, that deep ocean mineral water may improve exercise recovery, aerobic exercise performance, improve lower leg power output and hydration status compared to either placebo or sports drink. Furthermore, animal models support these plausibilities with improved mitochondrial biogenesis, biomolecules of exercises performance, cardiovascular hemodynamics, inflammatory cytokine responses to exercise and overall exercise adaptation.

As ocean minerals are absorbed by marine organisms, Algae species such as Lithothamnion have higher concentrations of the same ocean minerals but structured differently at the nano scale and thus may have the potential to be more effective at improving exercise phenotypes. Therefore, the proposed exploratory RCT will investigate the effects of water soluble Lithothamnion species on exhaustive exercise-induced lactate accumulation, recovery and power output in trained cyclists, compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male trained cyclist.
* Cycling for the purpose of exercise training (i.e. not cycling for transport) at least 100km per week for the last 6 months
* VȮ2peak that is greater than 50 ml˙kg˙ml-1

Exclusion Criteria:

* Any muscle disorder
* Serious medical co-morbidities
* Thyroid dysfunction or specific allergies
* Contraindications to dependent variables
* Currently participation in another research study
* Currently not talking other nutrition supplements

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Blood lactate concentration accumulation (measured using a Lactate Pro2 Portable Analyzer; Arkray, Tokyo, Japan) to repeated Wingate anaerobic exhaustive exercise performed on a Lode Excalibur cycle ergometer (Lode B.V., Groningen, DE). | 40 minute exercise protocol
  Pre, during and post repeated Wingate anaerobic exercise performance test (three Wingates separated by 3 minutes recovery) blood lactate accumulation (mmol/L) will be measured by capillary sampling and lactate recovery (mmol/L) will be measured for a subsequent 20 minutes. The primary outcome measure will be any difference in blood lactate response between the interventions after 7 days of supplementation with either Aqumin or a placebo (see arms and interventions section).

SECONDARY OUTCOMES:
Exercise performance via Wingate anaerobic exercise performance test for maximal power output (Watts) performed on a Lode Excalibur cycle ergometer (Lode B.V., Groningen, DE). | 40 minute exercise protocol.
  A repeated Wingate anaerobic exercise performance test (three Wingates separated by 3 minutes recovery) will be used to assessed pre and post intervention maximal lower-body power output (measured in absolute Watts (W) and relative power output (W/kg)) and fatigued power output (measured in absolute Watts (W) and relative power output (W/kg)). The secondary outcome measure will be any difference power output in response to 7 days of supplementation with either Aqumin or a placebo (see arms and interventions section).

CONTACTS AND LOCATIONS:
Overall Officials: Shane M Heffernan, PhD, Principal Investigator — University College Dublin; Katy Horner, PhD, Principal Investigator — University College Dublin

IPD SHARING:
Plan to Share IPD: Yes
All data and information will be presented in the peer reviewed manuscript.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the time of peer review publication.
Access Criteria: Peer review publication.

REFERENCES:
- [Background] Perez-Turpin JA, Trottini M, Chinchilla-Mira JJ, Cyganik W. Effects of seawater ingestion on lactate response to exercise in runners. Biol Sport. 2017 Dec;34(4):407-412. doi: 10.5114/biolsport.2017.70733. Epub 2017 Oct 10. PMID 29472745
- [Background] Fan H, Tan Z, Hua Y, Huang X, Gao Y, Wu Y, Liu B, Zhou Y. Deep sea water improves exercise and inhibits oxidative stress in a physical fatigue mouse model. Biomed Rep. 2016 Jun;4(6):751-757. doi: 10.3892/br.2016.651. Epub 2016 Apr 13. PMID 27284418
- [Background] Wei CY, Chen CY, Liao YH, Tsai YS, Huang CY, Chaunchaiyakul R, Higgins MF, Kuo CH. Deep Ocean Mineral Supplementation Enhances the Cerebral Hemodynamic Response during Exercise and Decreases Inflammation Postexercise in Men at Two Age Levels. Front Physiol. 2017 Dec 12;8:1016. doi: 10.3389/fphys.2017.01016. eCollection 2017. PMID 29311955
- [Background] Hou CW, Tsai YS, Jean WH, Chen CY, Ivy JL, Huang CY, Kuo CH. Deep ocean mineral water accelerates recovery from physical fatigue. J Int Soc Sports Nutr. 2013 Feb 12;10(1):7. doi: 10.1186/1550-2783-10-7. PMID 23402436
- [Background] Stasiule L, Capkauskiene S, Vizbaraite D, Stasiulis A. Deep mineral water accelerates recovery after dehydrating aerobic exercise: a randomized, double-blind, placebo-controlled crossover study. J Int Soc Sports Nutr. 2014 Jun 26;11:34. doi: 10.1186/1550-2783-11-34. eCollection 2014. PMID 25002835
- [Background] Keen DA, Constantopoulos E, Konhilas JP. The impact of post-exercise hydration with deep-ocean mineral water on rehydration and exercise performance. J Int Soc Sports Nutr. 2016 Apr 16;13:17. doi: 10.1186/s12970-016-0129-8. eCollection 2016. PMID 27087798
- [Background] Ha BG, Moon DS, Kim HJ, Shon YH. Magnesium and calcium-enriched deep-sea water promotes mitochondrial biogenesis by AMPK-activated signals pathway in 3T3-L1 preadipocytes. Biomed Pharmacother. 2016 Oct;83:477-484. doi: 10.1016/j.biopha.2016.07.009. Epub 2016 Jul 18. PMID 27434863
- [Background] Katsuda S, Yasukawa T, Nakagawa K, Miyake M, Yamasaki M, Katahira K, Mohri M, Shimizu T, Hazama A. Deep-sea water improves cardiovascular hemodynamics in Kurosawa and Kusanagi-Hypercholesterolemic (KHC) rabbits. Biol Pharm Bull. 2008 Jan;31(1):38-44. doi: 10.1248/bpb.31.38. PMID 18175939
- [Background] Saovieng S, Wu J, Huang CY, Kao CL, Higgins MF, Chuanchaiyakul R, Kuo CH. Deep Ocean Minerals Minimize Eccentric Exercise-Induced Inflammatory Response of Rat Skeletal Muscle. Front Physiol. 2018 Sep 28;9:1351. doi: 10.3389/fphys.2018.01351. eCollection 2018. PMID 30323766
- [Background] Wang, S.-T., Hwang, D.-F., Chen, R.-H., & Chen, Y.-C. (2009). Effect of deep sea water on the exercise-induced fatigue of rats. Journal of Food and Drug Analysis, 17(2), 133-141.
- [Background] Heffernan SM, Horner K, De Vito G, Conway GE. The Role of Mineral and Trace Element Supplementation in Exercise and Athletic Performance: A Systematic Review. Nutrients. 2019 Mar 24;11(3):696. doi: 10.3390/nu11030696. PMID 30909645